CLINICAL TRIAL: NCT00391014
Title: AMBINEB: Clinical Trial to Evaluate Tolerance and Safety of Nebulized Liposomal Amphotericin B Ambisome for Prophylaxis of Invasive Pulmonary Aspergillosis in Patients With Acute Myeloid Leukemia and Allogeneic Haematopoietic Progenitor Cell Transplant (Alo-HPCT)
Brief Title: Nebulized Liposomal Amphotericin B Ambisome for Prophylaxis of Invasive Pulmonary Aspergillosis
Acronym: AMBINEB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2005-000703-34; AMBINEB
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Acute Myeloid Leukemia; Allogeneic Haematopoietic Progenitor Cell Transplant
Keywords: Acute myeloid Leukemia; Allogeneic haematopoietic progenitor cell transplant; Acute Invasive Aspergillosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): AML patients in induction chemotherapy treatment will received prophylaxis with nebulized liposomal amphotericin B (24 mg/week). It will be maintained during the intensification chemotherapy and in periods between cycles.
  If patient required ALO-TPH, the prophylaxis should be followed.
  Interventions: Drug: liposomal Amphotericine B

INTERVENTIONS:
Drug: liposomal Amphotericine B — AML patients in induction chemotherapy treatment will received prophylaxis with nebulized liposomal amphotericin B (24 mg/week). It will be maintained during the intensification chemotherapy and in periods between cycles.
  If patient required ALO-TPH, the prophylaxis should be followed.

SUMMARY:
The trial is planned as a multicentric, national, phase II, open-label trial to evaluate safety and tolerance of nebulized Liposomal Amphotericin B (Ambisome) for LMA patients during the induction therapy ,intensification, plus Allogeneic Haematopoietic Progenitor Cell transplant in due course, as well for patients diagnosed of several malignant haematologic diseases and treated with Allogeneic Haematopoietic Progenitor Cell Transplant

DETAILED DESCRIPTION:
The invasive fungal infection (IFI) is the most common cause of mortality related to autologous stem cell transplant. Taking into account that Saprophytic Aspergillus is usually acquired by inhalation, to protect the bronchial tree just before the tissue invasion is quite attractive. In haematologic patients, as well as those ones subjected to an Allogeneic haematopoietic progenitor cell transplant, there is another group of patients at high risk of Invasive Pulmonary Aspergillosis (IPA). These are those patients with acute myeloid leucemia (AML), submitted to induction, intensification or consolidation polychemotherapy. The IPA incidence rate in these patients, whenever during their evolution, reaches 18-20%, with usual treatments. Furthermore, unlike allogeneic haematopoietic progenitor cell transplant patients, neutropenia was the only IPA risk factor. Nowadays, pharmacologic prophylaxis against IPA, in patients with allogeneic haematopoietic progenitor cell transplant and patients affected by AML in induction or intensification therapy is far from being optimal, because of problems related to tolerance and drug interactions .

The Nebulized Liposomal Amphotericin B (Ambisome) prophylaxis against IPA has shown good tolerance, safety and efficacy in lung transplant recipients.

Extrapolating the results obtained in lung transplant recipients, we get the conclusion that it would be essential to study safety and tolerance of nebulized AMBISOME in the group of patients with different peculiarities, mucositis secondary to chemotherapy, and high incidence of IPA in order to reach the goal of evaluate its efficacy as prophylaxis against IPA in this kind of patients

ELIGIBILITY:
Inclusion Criteria:

* Patient has decided voluntary to consent his or her participation signing the consent form before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patients with Acute myeloid Leukemia (AML), that will start induction chemotherapy or those patients submitted to an Allogeneic haematopoietic progenitor cell transplant.
* The patient is >18 years old.

Exclusion Criteria:

* Patient with prior Invasive Pulmonary Aspergillosis (IPA) history.
* History of allergy or hypersensitivity to Amphotericin B.
* Patient with intellectual deficit or patients with psychological alterations that make impossible the trial understanding.
* Pregnancy or breastfeeding.
* Patient has received other investigational drug or non traded product within 30 days before trial beginning.
* Patient is enrolled in another clinical research study or/and is receiving an investigational agent for any reason.
* Patient had major surgery within 4 weeks before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety prophylaxis against IPA in LMA patients. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ruiz Isabel, Dr, Principal Investigator — Hospital Vall d'Hebron; Rovira Montserrat, Dr, Principal Investigator — Hospital Clinic of Barcelona
Locations (4):
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital Universitario la Fe, Valencia, Valencia
  - Hospital Universitario de Salamanca, Salamanca

REFERENCES:
- [Background] Denning DW. Invasive aspergillosis. Clin Infect Dis. 1998 Apr;26(4):781-803; quiz 804-5. doi: 10.1086/513943. No abstract available. PMID 9564455
- [Background] Marr KA, Carter RA, Boeckh M, Martin P, Corey L. Invasive aspergillosis in allogeneic stem cell transplant recipients: changes in epidemiology and risk factors. Blood. 2002 Dec 15;100(13):4358-66. doi: 10.1182/blood-2002-05-1496. Epub 2002 Aug 22. PMID 12393425
- [Background] Winston DJ, Maziarz RT, Chandrasekar PH, Lazarus HM, Goldman M, Blumer JL, Leitz GJ, Territo MC. Intravenous and oral itraconazole versus intravenous and oral fluconazole for long-term antifungal prophylaxis in allogeneic hematopoietic stem-cell transplant recipients. A multicenter, randomized trial. Ann Intern Med. 2003 May 6;138(9):705-13. doi: 10.7326/0003-4819-138-9-200305060-00006. PMID 12729424
- [Background] Siwek GT, Dodgson KJ, de Magalhaes-Silverman M, Bartelt LA, Kilborn SB, Hoth PL, Diekema DJ, Pfaller MA. Invasive zygomycosis in hematopoietic stem cell transplant recipients receiving voriconazole prophylaxis. Clin Infect Dis. 2004 Aug 15;39(4):584-7. doi: 10.1086/422723. Epub 2004 Jul 30. PMID 15356827
- [Background] Kramer MR, Denning DW, Marshall SE, Ross DJ, Berry G, Lewiston NJ, Stevens DA, Theodore J. Ulcerative tracheobronchitis after lung transplantation. A new form of invasive aspergillosis. Am Rev Respir Dis. 1991 Sep;144(3 Pt 1):552-6. doi: 10.1164/ajrccm/144.3_Pt_1.552. PMID 1654038
- [Background] Yeldandi V, Laghi F, McCabe MA, Larson R, O'Keefe P, Husain A, Montoya A, Garrity ER Jr. Aspergillus and lung transplantation. J Heart Lung Transplant. 1995 Sep-Oct;14(5):883-90. PMID 8800724
- [Background] Westney GE, Kesten S, De Hoyos A, Chapparro C, Winton T, Maurer JR. Aspergillus infection in single and double lung transplant recipients. Transplantation. 1996 Mar 27;61(6):915-9. doi: 10.1097/00007890-199603270-00013. PMID 8623160
- [Background] Cahill BC, Hibbs JR, Savik K, Juni BA, Dosland BM, Edin-Stibbe C, Hertz MI. Aspergillus airway colonization and invasive disease after lung transplantation. Chest. 1997 Nov 5;112(5):1160-4. doi: 10.1378/chest.112.5.1160. PMID 9367451
- [Background] Reichenspurner H, Gamberg P, Nitschke M, Valantine H, Hunt S, Oyer PE, Reitz BA. Significant reduction in the number of fungal infections after lung-, heart-lung, and heart transplantation using aerosolized amphotericin B prophylaxis. Transplant Proc. 1997 Feb-Mar;29(1-2):627-8. doi: 10.1016/s0041-1345(96)00363-6. No abstract available. PMID 9123449
- [Background] Calvo V, Borro JM, Morales P, Morcillo A, Vicente R, Tarrazona V, Paris F. Antifungal prophylaxis during the early postoperative period of lung transplantation. Valencia Lung Transplant Group. Chest. 1999 May;115(5):1301-4. doi: 10.1378/chest.115.5.1301. PMID 10334143
- [Background] Dubois J, Bartter T, Gryn J, Pratter MR. The physiologic effects of inhaled amphotericin B. Chest. 1995 Sep;108(3):750-3. doi: 10.1378/chest.108.3.750. PMID 7656628
- [Background] Schmitt HJ, Bernard EM, Hauser M, Armstrong D. Aerosol amphotericin B is effective for prophylaxis and therapy in a rat model of pulmonary aspergillosis. Antimicrob Agents Chemother. 1988 Nov;32(11):1676-9. doi: 10.1128/AAC.32.11.1676. PMID 3252750
- [Background] Monforte V, Roman A, Gavalda J, Bravo C, Tenorio L, Ferrer A, Maestre J, Morell F. Nebulized amphotericin B prophylaxis for Aspergillus infection in lung transplantation: study of risk factors. J Heart Lung Transplant. 2001 Dec;20(12):1274-81. doi: 10.1016/s1053-2498(01)00364-3. PMID 11744410
- [Background] Monforte V, Roman A, Gavalda J, Lopez R, Pou L, Simo M, Aguade S, Soriano B, Bravo C, Morell F. Nebulized amphotericin B concentration and distribution in the respiratory tract of lung-transplanted patients. Transplantation. 2003 May 15;75(9):1571-4. doi: 10.1097/01.TP.0000054233.60100.7A. PMID 12792517
- [Background] Lambros MP, Bourne DW, Abbas SA, Johnson DL. Disposition of aerosolized liposomal amphotericin B. J Pharm Sci. 1997 Sep;86(9):1066-9. doi: 10.1021/js9604218. PMID 9294824
- [Background] Thomas DA, Myers MA, Wichert B, Schreier H, Gonzalez-Rothi RJ. Acute effects of liposome aerosol inhalation on pulmonary function in healthy human volunteers. Chest. 1991 May;99(5):1268-70. doi: 10.1378/chest.99.5.1268. PMID 2019191
- [Background] Kume H, Yamazaki T, Abe M, Tanuma H, Okudaira M, Okayasu I. Increase in aspergillosis and severe mycotic infection in patients with leukemia and MDS: comparison of the data from the Annual of the Pathological Autopsy Cases in Japan in 1989, 1993 and 1997. Pathol Int. 2003 Nov;53(11):744-50. doi: 10.1046/j.1440-1827.2003.01548.x. PMID 14629297
- [Background] Nosari A, Oreste P, Cairoli R, Montillo M, Carrafiello G, Astolfi A, Muti G, Marbello L, Tedeschi A, Magliano E, Morra E. Invasive aspergillosis in haematological malignancies: clinical findings and management for intensive chemotherapy completion. Am J Hematol. 2001 Dec;68(4):231-6. doi: 10.1002/ajh.1187. PMID 11754411
- [Background] Behre GF, Schwartz S, Lenz K, Ludwig WD, Wandt H, Schilling E, Heinemann V, Link H, Trittin A, Boenisch O, et al. Aerosol amphotericin B inhalations for prevention of invasive pulmonary aspergillosis in neutropenic cancer patients. Ann Hematol. 1995 Dec;71(6):287-91. doi: 10.1007/BF01697981. PMID 8534760
- [Background] Schwartz S, Behre G, Heinemann V, Wandt H, Schilling E, Arning M, Trittin A, Kern WV, Boenisch O, Bosse D, Lenz K, Ludwig WD, Hiddemann W, Siegert W, Beyer J. Aerosolized amphotericin B inhalations as prophylaxis of invasive aspergillus infections during prolonged neutropenia: results of a prospective randomized multicenter trial. Blood. 1999 Jun 1;93(11):3654-61. PMID 10339471
- [Background] Conneally E, Cafferkey MT, Daly PA, Keane CT, McCann SR. Nebulized amphotericin B as prophylaxis against invasive aspergillosis in granulocytopenic patients. Bone Marrow Transplant. 1990 Jun;5(6):403-6. PMID 2196098
- [Background] Myers SE, Devine SM, Topper RL, Ondrey M, Chandler C, O'Toole K, Williams SF, Larson RA, Geller RB. A pilot study of prophylactic aerosolized amphotericin B in patients at risk for prolonged neutropenia. Leuk Lymphoma. 1992 Oct;8(3):229-33. doi: 10.3109/10428199209054909. PMID 1490149
- [Background] Erjavec Z, Woolthuis GM, de Vries-Hospers HG, Sluiter WJ, Daenen SM, de Pauw B, Halie MR. Tolerance and efficacy of Amphotericin B inhalations for prevention of invasive pulmonary aspergillosis in haematological patients. Eur J Clin Microbiol Infect Dis. 1997 May;16(5):364-8. doi: 10.1007/BF01726364. PMID 9228476
- [Background] Hertenstein B, Kern WV, Schmeiser T, Stefanic M, Bunjes D, Wiesneth M, Novotny J, Heimpel H, Arnold R. Low incidence of invasive fungal infections after bone marrow transplantation in patients receiving amphotericin B inhalations during neutropenia. Ann Hematol. 1994 Jan;68(1):21-6. doi: 10.1007/BF01695915. PMID 8110874
- See also: Spanish association of Haematology — http://www.aehh.org